CLINICAL TRIAL: NCT06073197
Title: Comparision of the Effects of Ultrasound-guided Erector Spinae Block and Combined Deep and Superficial Serratus Anterior Plane Block on Perioperative Analgesia for Video-assisted Thoracoscopic Surgery.
Brief Title: Comparison of Erector Spinae Block and Combined Deep and Superficial Serratus Anterior Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Seda Cansabuncu, medical doctor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-11/19
Record Dates: First submitted 2023-09-19; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Analgesia; Pain, Postoperative; Thoracic; Anesthesia
Keywords: serratus anterior plane block; video-assisted thoracoscopic surgery; erector spinae block; postoperative analgesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: randomized, controlled
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erector spinae plane block (Active Comparator): Plane blocks implemented on preoperative course on 35 patients for group.
  Interventions: Procedure: erector spinae plane block
- combined deep and superficial serratus anterior plane block (Active Comparator): Plane blocks implemented on preoperative course on 35 patients for group.
  Interventions: Procedure: combined deep and superficial serratus anterior plane block

INTERVENTIONS:
Procedure: erector spinae plane block — Erector spinae plane block was implemented on preoperative course on 35 patients. Intraoperative analgesic (Fentanyl) consumption was measured for intraoperative effects of the erector spinae plane block. Postoperative Visual Analogue Scale (VAS, from 0 to 10) scores and postoperative analgesic (Morphine) consumption was measured using Mann-Whitney test.
  Arms: erector spinae plane block
Procedure: combined deep and superficial serratus anterior plane block — Combined deep and superficial serratus anterior plane block was implemented on preoperative course on 35 patients. Intraoperative analgesic (Fentanyl) consumption was measured for intraoperative effects of the erector spinae plane block Postoperative Visual Analogue Scale (VAS, from 0 to 10) scores and postoperative analgesic (Morphine) consumption was measured using Mann-Whitney test.
  Arms: combined deep and superficial serratus anterior plane block

SUMMARY:
Objective: The authors hypothesized that combined deep and superficial serratus anterior plane block (SAPB) is as effective as erector spinae plane block (ESPB) for intraoperative and postoperative analgesia for video-assisted thoracoscopic surgery.

Design: A prospective randomized controlled study. Participants: Adult patients undergoing elective video-assisted thoracoscopic surgery.

Interventions: Preoperative SAPB or ESPB implementation.

DETAILED DESCRIPTION:
Plane blocks implemented on preoperative course on 35 patients for each group. Postoperative Visual Analogue Scale (VAS) scores (0-10), intraoperative and postoperative analgesic consumption was measured using Mann-Whitney test. In the postoperative phase, opioid side effects, complications related to plane blocks, mobilization time and length of hospital stay was recorded and measured.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) classification I-II scheduled for elective VATS

Exclusion Criteria:

* Patients who did not give consent
* Local anaesthetic allergy
* Known or suspected coagulopathy
* İnfection at the injection site
* History of thoracic surgery
* Severe cardiovascular disease
* Hepatic or renal insufficiency (glomerular filtration rate <15 ml/min/1.73 m2)
* Severe neurological or psychiatric disorders
* Chronic opioid use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
postoperative analgesic effects | first 48 hours
  The primary outcome is compare the postoperative analgesic effects of SAPB and ESPB applied under USG guidance before surgery in patients scheduled for VATS using VAS (Visual Analogue Scale from 0 to 10).
intraoperative analgesic effects | intraoperative phase
  The primary outcome is compare the intraoperative analgesic effects of SAPB and ESPB applied under USG guidance before surgery in patients scheduled for VATS by measuring perioperative fentanyl consumption in both groups.

SECONDARY OUTCOMES:
side effects | first 48 hours
  The secondary aim was to compare the opioid side effects. Patients were informed about opioid side effects and asked whether side effects were present.
complications | first 48 hours
  The secondary aim was to compare the complications related to the applied block. Patients were examined and evaluated for any complications related to the block.
mobilization | first 48 hours
  The secondary aim was to compare the mobilization time
stay of hospital | first 4 days
  length of stay in the recovery unit and hospital

CONTACTS AND LOCATIONS:
Overall Officials: seda cansabuncu, Study Chair — Uludag University
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)